CLINICAL TRIAL: NCT00644787
Title: A Phase II/III Study of JNS020QD in Cancer Pain Patients - A Dose-Finding, Double-Blind Study of JNS020QD Compared With JNS005 in Patients Previously Untreated With Opioid Analgesics
Brief Title: A Dose-Finding Study of Fentanyl (JNS020 QD) 1-Day Transdermal Patch in Participants With Cancer Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014899; JNS020QD-JPN-C02
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Pain; Cancer
Keywords: Pain; Cancer; Fentanyl; JNS020QD; JNS005
MeSH Terms: conditions — Pain; Neoplasms | interventions — Fentanyl; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fentanyl 1-day transdermal patch (Titration Phase) (Experimental): Fentanyl 1-day application transdermal patch releasing the drug at the rate of 12.5 microgram per hour (mcg/hr) applied once daily, and maintained for 2 days. Dose escalation or reduction is done as per Investigator's discretion (maximum applied dose is 100 mcg/hr) up to Day 11 and then dose is fixed up to end of treatment period, that is Day 14. Participants who met the predefined criteria at the end of Titration Phase enter the Double Blind Phase.
  Interventions: Drug: Fentanyl 1-day transdermal patch (Titration Phase)
- Fentanyl 1-day transdermal patch (Double Blind Phase) (Experimental): Participants who meet the predefined criteria at the end of Titration Phase and enter the Double Blind Phase receive fentanyl 1-day application transdermal patch and placebo matched to fentanyl 3-day application (JNS005) transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
  Interventions: Drug: Fentanyl 1-day transdermal patch (Double Blind Phase); Drug: Placebo
- Fentanyl 3-day transdermal patch (Double Blind Phase) (Active Comparator): Participants who meet the predefined criteria at the end of Titration Phase and enter the Double Blind Phase receive fentanyl 3-day application transdermal patch and placebo matched to fentanyl 1-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
  Interventions: Drug: Fentanyl 3-day transdermal patch (Double Blind Phase); Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl 1-day transdermal patch (Titration Phase) — Fentanyl 1-day application transdermal patch releasing the drug at the rate of 12.5 mcg/hr applied once daily, and maintained for 2 days. Dose escalation or reduction is done as per Investigator's discretion (maximum applied dose is 100 mcg/hr) up to Day 11 and then dose is fixed up to end of treatment period, that is Day 14.
  Other Names: JNS020QD
  Arms: Fentanyl 1-day transdermal patch (Titration Phase)
Drug: Fentanyl 1-day transdermal patch (Double Blind Phase) — Fentanyl 1-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
  Other Names: JNS020QD
  Arms: Fentanyl 1-day transdermal patch (Double Blind Phase)
Drug: Fentanyl 3-day transdermal patch (Double Blind Phase) — Fentanyl 3-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
  Other Names: JNS005
  Arms: Fentanyl 3-day transdermal patch (Double Blind Phase)
Drug: Placebo — Placebo matching to fentanyl 3-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase for 10 days.
  Arms: Fentanyl 1-day transdermal patch (Double Blind Phase)
Drug: Placebo — Placebo matching to fentanyl 1-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase for 10 days.
  Arms: Fentanyl 3-day transdermal patch (Double Blind Phase)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fentanyl 1-day application (JNS020QD) transdermal patch (patch containing a drug that is put on the skin so the drug can enter the body through the skin) and to assess the non-inferiority of fentanyl 1-day application transdermal patch to fentanyl 3-day application (JNS005) transdermal patch in participants with cancer pain.

DETAILED DESCRIPTION:
This is a multi-center (conducted in more than one center) study, consisting of two periods: Period 1 is open-label (all people know the identity of the intervention), non-comparative dose titration phase and Period 2 is double blind (neither physician nor participant knows the treatment that the participant receives), positive control (fentanyl 3-day application transdermal patch is used as control drug) phase. In Period 1, fentanyl 1-day application transdermal patch 12.5 microgram per hour (mcg/hr) will be applied to chest, abdomen, upper arm or thigh and will be maintained for 2 days to ensure the safety of participants. Dose escalation or reduction will be allowed based on participant's condition from Day 3 to Day 11 and thereafter dose will be maintained from Day 11 to Day 13 with a maximum application dose of 100 mcg/hr. The total duration of Period 1 is 14 days (a total of 13 applications; including the day of final patch removal). Participants who met the predefined criteria at the end of dose titration phase will enter the double blind phase. In double blind phase, participants will receive either fentanyl 1-day application transdermal patch and placebo matched to fentanyl 3-day application transdermal patch or fentanyl 3-day application transdermal patch and placebo matched to fentanyl 1-day application transdermal patch at the same dose as used at the completion of Period 1. The duration of Period 2 is 10 days. Efficacy will primarily be evaluated by percentage of participants achieving dose titration success and change in mean visual analog scale (VAS) score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cancer pain who were previously not treated with opioid analgesics (drug used to control pain)
* Participants with a pain score of greater than or equal to 35 millimeter (mm) on a 100-mm visual analog scale (VAS)
* Participants who are considered to have "insufficient response" to non-opioid analgesics and require treatment with opioid analgesics by the physician
* Participants who have an established diagnosis of cancer and are notified of the disease
* Participants who can be hospitalized during Period 1 (dose-titration period)

Exclusion Criteria:

* Participants with impaired respiratory function due to chronic lung disease or others
* Participants with asthma (breathing disorder in which there is wheezing and difficulty in breathing)
* Participants with bradyarrhythmia (slow, irregular heartbeats)
* Participants with following measurements indicative of hepatic or renal impairment during the pre-treatment observation period: Aspartate transaminase (AST) greater than 5 times the upper limit of reference range, Alanine transaminase (ALT) greater than 5 times the upper limit of reference range, serum creatinine greater than 3 times the upper limit of reference range
* Participants with any cerebral damage, such as brain tumor, accompanied by increased intracranial pressure, disturbance of consciousness, coma, or respiratory disturbance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (43):
- Japan (43):
  - Asahi
  - Asahikawa
  - Bunkyō City
  - Chiba
  - Chikushino-shi
  - Fukuoka
  - Fushimi
  - Higashi-Ibaraki
  - Himeji
  - Hirosaki
  - Hiroshima
  - Hitachi
  - Hohfu
  - Ichinomiya
  - Ikeda
  - Iwakuni
  - Kawachi-Nagano
  - Kawasaki
  - Kitakyushu
  - Kiyose
  - Kobe
  - Kochi
  - Matsue
  - Matsuyama
  - Nishinomiya
  - Okayama
  - Osaka
  - Ōita
  - Ōtake
  - Sakai
  - Sendai
  - Shigenobu N/A
  - Sonogishukugō
  - Sunto
  - Tamaho N/A
  - Tokushima
  - Tokyo
  - Toyohashi
  - Tsukuba
  - Utsunomiya
  - Wako
  - Yamaguchi
  - Yonago

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl 1-day Transdermal Patch (Titration Phase): Fentanyl 1-day application (JNS020QD) transdermal patch (patch containing a drug that was put on skin so the drug entered the body through the skin) releasing the drug at the rate of 12.5 microgram per hour (mcg/hr) applied once daily, and maintained for 2 days. Dose escalation or reduction was done as per Investigator's discretion (maximum applied dose was 100 mcg/hr) up to Day 11 and then dose was fixed up to end of treatment period, that is Day 14. Participants who met the predefined criteria at the end of Titration Phase entered the Double Blind Phase.
- Fentanyl 1-day Transdermal Patch (Double Blind Phase): Participants who met the predefined criteria at the end of Titration Phase and entered the Double Blind Phase received fentanyl 1-day application transdermal patch and placebo matched to fentanyl 3-day application (JNS005) transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
- Fentanyl 3-day Transdermal Patch (Double Blind Phase): Participants who met the predefined criteria at the end of Titration Phase and entered the Double Blind Phase received fentanyl 3-day application transdermal patch and placebo matched to fentanyl 1-day application transdermal patch applied once daily releasing the drug at the same dose as maintained at the end of Titration Phase with maximum applied dose of 100 mcg/hr for 10 days.
Period: Period 1: Titration Phase
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase) | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Started | 156 | 0 | 0
Completed | 129 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Worsening of underlying disease | 5 | 0 | 0
Not completed — Worsening of complications | 1 | 0 | 0
Not completed — Worsening of symptoms | 1 | 0 | 0
Not completed — Dose adjustment required on Day 12 or 13 | 3 | 0 | 0
Not completed — Participant was judged as ineligible | 3 | 0 | 0
Period: Period 2: Double Blind Phase
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase) | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Started | 0 | 58 | 62
Completed | 0 | 49 | 55
Not Completed | 0 | 9 | 7
Not completed — Adverse Event | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Worsening of underlying disease | 0 | 6 | 2
Not completed — Worsening of symptoms | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Out of a total of 156 participants, Baseline characteristics were available for only 155 participants who were included in Full Analysis Set (FAS) population. FAS population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug.
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Dose Titration Success
Description: Participants achieving dose titration success included all participants who had a mean Visual Analog Scale (VAS) score of less than or equal to 34 millimeter (mm) and received not more than 2 rescue doses during the last 3 days before the completion or discontinuation of dose titration phase. Pain Intensity VAS measured severity of pain on a 100 mm scale ranging from 0 mm (no pain) to 100 mm (severest pain conceivable) and rescue dose was defined as dose of a fast-acting oral morphine hydrochloride solution or morphine in water solution used in the case of breakthrough pain.
Time Frame: Day 14 or early discontinuation (ED)
Population: Full Analysis Set (FAS) population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Percentage of participants | 80.60 [73.50 to 86.50]

2. Primary Outcome: Change From Dose Titration Phase in the Mean Visual Analog Scale (VAS) Score at Double Blind Phase
Description: The mean VAS score for the last 3 days before the completion or discontinuation of Double Blind Phase was compared with that for the last 3 days before the completion or discontinuation of Dose Titration Phase and the change from Dose Titration Phase in the mean VAS Score at Double Blind Phase was reported. Pain Intensity VAS measured severity of pain on a 100 mm scale ranging from 0 mm (no pain) to 100 mm (severest pain conceivable).
Time Frame: Dose Titration Phase (Day 12 to Day 14) and Double Blind Phase (Day 8 to Day 10)
Population: Per Protocol Set (PPS) population included all the participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug excluding those with any major protocol deviation or other violations.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
mm
  Dose Titration Phase (Day 12 to Day 14) | 18.4 (9.05) | 20.6 (8.58)
  Change at Double Blind Phase (Day 8 to Day 10) | -1.1 (14.82) | -2.5 (11.32)
Statistical Analysis 1: Comparison: Fentanyl 1-day Transdermal Patch (Double Blind Phase) vs Fentanyl 3-day Transdermal Patch (Double Blind Phase); Test type: Non-Inferiority or Equivalence — Difference of 7.5 mm in VAS score was selected as the threshold value for clinical non-inferiority of Fentanyl 1-day transdermal patch to Fentanyl 3-day transdermal patch; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-3.50 to 6.23]

3. Secondary Outcome: Number of Participants With Response Based on Participant's Global Assessment Scale in Titration Phase
Description: Participants were asked to assess their satisfaction with respect to the therapeutic efficacy (effectiveness) of the study drug to control pain on a 5-point scale ranging from 1 to 5, where 1 = extremely satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied and 5 = extremely dissatisfied.
Time Frame: Day 1 pre-application (PA), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13 and Day 14 or ED
Population: The FAS population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Participants
  Day 1 PA; Extremely satisfied (n=155) | 1 [3.10 to 11.50]
  Day 1 PA; Satisfied (n=155) | 9 [50.50 to 66.50]
  Day1 PA;Neither satisfied nor dissatisfied(n=155) | 54
  Day 1 PA; Dissatisfied (n=155) | 83
  Day 1 PA; Extremely dissatisfied (n=155) | 8
  Day 2; Extremely satisfied (n=155) | 4
  Day 2; Satisfied (n=155) | 32
  Day 2; Neither satisfied nor dissatisfied (n=155) | 79
  Day 2; Dissatisfied (n=155) | 39
  Day 2; Extremely dissatisfied (n=155) | 1
  Day 3; Extremely satisfied (n=153) | 1
  Day 3; Satisfied (n=153) | 50
  Day 3; Neither satisfied nor dissatisfied (n=153) | 70
  Day 3; Dissatisfied (n=153) | 31
  Day 3; Extremely dissatisfied (n=153) | 1
  Day 4; Extremely satisfied (n=152) | 3
  Day 4; Satisfied (n=152) | 55
  Day 4; Neither satisfied nor dissatisfied (n=152) | 69
  Day 4; Dissatisfied (n=152) | 24
  Day 4; Extremely dissatisfied (n=152) | 1
  Day 5; Extremely satisfied (n=151) | 4
  Day 5; Satisfied (n=151) | 63
  Day 5; Neither satisfied nor dissatisfied (n=151) | 59
  Day 5; Dissatisfied (n=151) | 24
  Day 5; Extremely dissatisfied (n=151) | 1
  Day 6; Extremely satisfied (n=129) | 4
  Day 6; Dissatisfied (n=129) | 54
  Day 6; Extremely dissatisfied (n=129) | 51
  Day 6; Satisfied (n=129) | 19
  Day 6; Neither satisfied nor dissatisfied (n=129) | 1
  Day 7; Extremely satisfied (n=112) | 5
  Day 7; Satisfied (n=112) | 50
  Day 7; Neither satisfied nor dissatisfied (n=112) | 43
  Day 7; Dissatisfied (n=112) | 14
  Day 7; Extremely dissatisfied (n=112) | 0
  Day 8; Extremely satisfied (n=98) | 3
  Day 8; Satisfied (n=98) | 48
  Day 8; Neither satisfied nor dissatisfied (n=98) | 38
  Day 8; Dissatisfied (n=98) | 9
  Day 8; Extremely dissatisfied (n=98) | 0
  Day 9; Extremely satisfied (n=74) | 1
  Day 9; Satisfied (n=74) | 36
  Day 9; Neither satisfied nor dissatisfied (n=74) | 33
  Day 9; Dissatisfied (n=74) | 4
  Day 9; Extremely dissatisfied (n=74) | 0
  Day 10; Extremely satisfied (n=57) | 0
  Day 10; Satisfied (n=57) | 29
  Day 10; Neither satisfied nor dissatisfied (n=57) | 23
  Day 10; Dissatisfied (n=57) | 5
  Day 10; Extremely dissatisfied (n=57) | 0
  Day 11; Extremely satisfied (n=51) | 1
  Day 11; Satisfied (n=51) | 23
  Day 11; Neither satisfied nor dissatisfied (n=51) | 21
  Day 11; Dissatisfied (n=51) | 6
  Day 11; Extremely dissatisfied (n=51) | 0
  Day 12; Extremely satisfied (n=38) | 1
  Day 12; Satisfied (n=38) | 20
  Day 12; Neither satisfied nor dissatisfied (n=38) | 15
  Day 12; Dissatisfied (n=38) | 2
  Day 12; Extremely dissatisfied (n=38) | 0
  Day 13; Extremely satisfied (n=29) | 0
  Day 13; Satisfied (n=29) | 18
  Day 13; Neither satisfied nor dissatisfied (n=29) | 9
  Day 13; Dissatisfied (n=29) | 2
  Day 13; Extremely dissatisfied (n=29) | 0
  Day 14/ED; Extremely satisfied (n=155) | 9
  Day 14/ED; Satisfied (n=155) | 82
  Day14/ED;Neither satisfied nor dissatisfied(n=155) | 53
  Day 14/ED; Dissatisfied (n=155) | 11
  Day 14/ED; Extremely dissatisfied (n=155) | 0

4. Secondary Outcome: Number of Participants With Response Based on Participant's Global Assessment Scale in Double Blind Phase
Description: Participants were asked to assess their satisfaction with respect to the therapeutic efficacy of the study drug to control pain on a 5-point scale ranging from 1 to 5, where 1 = extremely satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied and 5 = extremely dissatisfied.
Time Frame: Day 14-End of Titration Phase (ETP), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9 and Day 10 or ED
Population: The PPS population included all the participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug excluding those with any major protocol deviation or other violations. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
Participants
  ETP; Extremely satisfied (n=54,60) | 3 [48.70 to 75.70] | 4 [55.00 to 79.70]
  ETP; Satisfied (n=54,60) | 31 [50.60 to 77.30] | 37 [46.50 to 72.40]
  ETP;Neither satisfied nor dissatisfied(n=54,60) | 19 | 16
  ETP; Dissatisfied (n=54,60) | 1 | 3
  Day 2; Extremely satisfied (n=54,60) | 3 | 4
  Day 2; Satisfied (n=54,60) | 33 | 38
  Day 2;Neither satisfied nor dissatisfied(n=54,60) | 16 | 16
  Day 2; Dissatisfied (n=54,60) | 2 | 2
  Day 3; Extremely satisfied (n=54,60) | 3 | 4
  Day 3; Satisfied (n=54,60) | 32 | 39
  Day 3;Neither satisfied nor dissatisfied(n=54,60) | 16 | 12
  Day 3; Dissatisfied (n=54,60) | 3 | 5
  Day 4; Extremely satisfied (n=54,60) | 3 | 5
  Day 4; Satisfied (n=54,60) | 31 | 33
  Day 4;Neither satisfied nor dissatisfied(n=54,60) | 17 | 19
  Day 4; Dissatisfied (n=54,60) | 3 | 3
  Day 5; Extremely satisfied (n=51,60) | 5 | 4
  Day 5; Satisfied (n=51,60) | 28 | 36
  Day 5;Neither satisfied nor dissatisfied(n=51,60) | 17 | 16
  Day 5; Dissatisfied (n=51,60) | 1 | 4
  Day 6; Extremely satisfied (n=50,60) | 6 | 6
  Day 6; Satisfied (n=50,60) | 25 | 34
  Day 6;Neither satisfied nor dissatisfied(n=50,60) | 17 | 15
  Day 6; Dissatisfied (n=50,60) | 2 | 5
  Day 7; Extremely satisfied (n=50,59) | 5 | 4
  Day 7; Satisfied (n=50,59) | 27 | 35
  Day 7;Neither satisfied nor dissatisfied(n=50,59) | 18 | 14
  Day 7; Dissatisfied (n=50,59) | 0 | 6
  Day 8; Extremely satisfied (n=50,59) | 5 | 4
  Day 8; Satisfied (n=50,59) | 25 | 31
  Day 8;Neither satisfied nor dissatisfied(n=50,59) | 19 | 17
  Day 8; Dissatisfied (n=50,59) | 1 | 7
  Day 9; Extremely satisfied (n=49,56) | 6 | 8
  Day 9; Satisfied (n=49,56) | 22 | 25
  Day 9;Neither satisfied nor dissatisfied(n=49,56) | 21 | 16
  Day 9; Dissatisfied (n=49,56) | 0 | 7
  Day 10/ED; Extremely satisfied (n=54,60) | 6 | 3
  Day 10/ED; Satisfied (n=54,60) | 29 | 33
  Day10/EDNeither satisfied nor dissatisfied;n=54,60 | 18 | 17
  Day 10/ED; Dissatisfied (n=54,60) | 1 | 7

5. Secondary Outcome: Pain Intensity Visual Analog Scale (VAS) Score in Titration Phase
Description: Participants were asked to assess their resting pain intensity (severity of pain) on a 100-mm VAS with the left edge (0 mm) defined as "no pain" and the right edge (100 mm) defined as "severest pain conceivable".
Time Frame: Day 1 PA, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13 and Day 14 or ED
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
mm
  Day 1 PA (n=155) | 56.8 (16.28)
  Day 2 (n=155) | 45.0 (18.93)
  Day 3 (n=153) | 41.9 (22.11)
  Day 4 (n=152) | 35.7 (19.43)
  Day 5 (n=151) | 32.7 (18.25)
  Day 6 (n=129) | 32.8 (19.15)
  Day 7 (n=111) | 30.5 (15.92)
  Day 8 (n=98) | 29.2 (15.40)
  Day 9 (n=74) | 29.0 (15.60)
  Day 10 (n=57) | 28.5 (15.35)
  Day 11 (n=51) | 25.8 (15.34)
  Day 12 (n=38) | 27.4 (17.93)
  Day 13 (n=29) | 27.5 (16.34)
  Day 14 or ED (n=155) | 23.8 (17.57)

6. Secondary Outcome: Pain Intensity Visual Analog Scale (VAS) Score in Double Blind Phase
Description: as for outcome 5
Time Frame: Day 14-End of Titration Phase (ETP), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9 and Day 10 or ED
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
mm
  ETP; (n=54,60) | 16.5 (9.34) | 18.6 (9.88)
  Day 2; (n=54,60) | 18.2 (11.31) | 18.4 (10.68)
  Day 3; (n=54,60) | 21.5 (19.56) | 17.8 (10.15)
  Day 4; (n=54,60) | 17.2 (14.09) | 18.5 (12.37)
  Day 5; (n=51,60) | 16.8 (14.43) | 17.7 (11.95)
  Day 6; (n=50,60) | 18.1 (16.08) | 19.2 (12.88)
  Day 7; (n=50,59) | 16.3 (14.33) | 18.0 (13.03)
  Day 8; (n=50,59) | 17.5 (16.71) | 17.2 (12.29)
  Day 9; (n=49,56) | 17.0 (18.10) | 17.2 (11.97)
  Day 10 or ED; (n=54,60) | 16.1 (16.10) | 18.8 (15.70)

7. Secondary Outcome: Percentage of Participants Achieving Pain Control in Double Blind Phase
Description: Pain control was assessed based on change in VAS and number of daily rescue doses during 3 days before completion of Double Blind Phase from 3 days before start of Double Blind Phase. For VAS score, difference of less than or equal to +15 mm and for rescue doses, difference of less than or equal to 1 was considered significant to achieve pain control. Pain Intensity VAS measured pain severity on a scale ranging from 0 mm (no pain) to 100 mm (severest pain conceivable) and rescue dose was defined as dose of fast-acting oral morphine formulation used in case of breakthrough pain.
Time Frame: Day 10 or ED
Population: The PPS population included all the participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug excluding those with any major protocol deviation or other violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
Percentage of participants | 83.3 [70.7 to 92.1] | 90.0 [79.5 to 96.2]

8. Secondary Outcome: Number of Participants With Pain Intensity Assessed by Categorical Scale for Pain in Titration Phase
Description: Participants were asked to assess their resting pain intensity (severity of pain) on a 4-point categorical scale ranging from 0 to 3 where 0 = no pain, 1 = mild pain, 2 = moderate pain and 3 = severe pain.
Time Frame: Day 1 PA, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13 and Day 14 or ED
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Participants
  Day 1 PA; No pain (n=155) | 0
  Day 1 PA; Mild pain (n=155) | 23
  Day 1 PA; moderate Pain (n=155) | 115
  Day 1 PA; severe Pain (n=155) | 17
  Day 2; No pain (n=155) | 4
  Day 2; Mild pain (n=155) | 54
  Day 2; Moderate pain (n=155) | 93
  Day 2; Severe pain (n=155) | 4
  Day 3; No pain (n=153) | 13
  Day 3; Mild pain (n=153) | 64
  Day 3; Moderate pain (n=153) | 69
  Day 3; Severe pain (n=153) | 7
  Day 4; No pain (n=152) | 12
  Day 4; Mild pain (n=152) | 68
  Day 4; Moderate pain (n=152) | 70
  Day 4; Severe pain (n=152) | 2
  Day 5; No pain (n=151) | 15
  Day 5; Mild pain (n=151) | 80
  Day 5; Moderate pain (n=151) | 50
  Day 5; Severe pain (n=151) | 6
  Day 6; No pain (n=129) | 13
  Day 6; Mild pain (n=129) | 69
  Day 6; Moderate pain (n=129) | 44
  Day 6; Severe pain (n=129) | 3
  Day 7; No pain (n=112) | 11
  Day 7; Mild pain (n=112) | 62
  Day 7; Moderate pain (n=112) | 36
  Day 7; Severe pain (n=112) | 3
  Day 8; No pain (n=98) | 9
  Day 8; Mild pain (n=98) | 56
  Day 8; Moderate pain (n=98) | 28
  Day 8; Severe pain (n=98) | 5
  Day 9; No pain (n=74) | 7
  Day 9; Mild pain (n=74) | 45
  Day 9; Moderate pain (n=74) | 22
  Day 9; Severe pain (n=74) | 0
  Day 10; No pain (n=57) | 3
  Day 10; Mild pain (n=57) | 31
  Day 10; Moderate pain (n=57) | 23
  Day 10; Severe pain (n=57) | 0
  Day 11; No pain (n=51) | 5
  Day 11; Mild pain (n=51) | 27
  Day 11; Moderate pain (n=51) | 18
  Day 11; Severe pain (n=51) | 1
  Day 12; No pain (n=38) | 5
  Day 12; Mild pain (n=38) | 21
  Day 12; Moderate pain (n=38) | 11
  Day 12; Severe pain (n=38) | 1
  Day 13; No pain (n=29) | 2
  Day 13; Mild pain (n=29) | 15
  Day 13; Moderate pain (n=29) | 12
  Day 13; Severe pain (n=29) | 0
  Day 14 or ED; No pain (n=155) | 20
  Day 14 or ED; Mild pain (n=155) | 92
  Day 14 or ED; Moderate pain(n=155) | 38
  Day 14 or ED; Severe pain(n=155) | 5

9. Secondary Outcome: Number of Participants With Pain Intensity Assessed by Categorical Scale for Pain in Double Blind Phase
Description: as for outcome 8
Time Frame: Day 14-End of Titration Phase (ETP), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9 and Day 10 or ED
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
Participants
  ETP; No pain (n=54,60) | 6 | 10
  ETP; MIld pain (n=54,60) | 39 | 37
  ETP; Moderate pain (n=54,60) | 9 | 12
  ETP; Severe pain (n=54,60) | 0 | 1
  Day 2; No pain (n=54,60) | 10 | 9
  Day 2; Mild pain (n=54,60) | 30 | 40
  Day 2; Moderate pain (n=54,60) | 14 | 11
  Day 2; Severe pain (n=54,60) | 0 | 0
  Day 3; No pain (n=54,60) | 9 | 12
  Day 3; Mild pain (n=54,60) | 34 | 39
  Day 3; Moderate pain (n=54,60) | 9 | 8
  Day 3; Severe pain (n=54,60) | 2 | 1
  Day 4; No pain (n=54,60) | 8 | 12
  Day 4; Mild pain (n=54,60) | 36 | 41
  Day 4; Moderate pain (n=54,60) | 10 | 7
  Day 4; Severe pain (n=54,60) | 0 | 0
  Day 5; No pain (n=51,60) | 8 | 11
  Day 5; Mild pain (n=51,60) | 31 | 42
  Day 5; Moderate pain (n=51,60) | 11 | 7
  Day 5; Severe pain (n=51,60) | 1 | 0
  Day 6; No pain (n=50,60) | 10 | 11
  Day 6; Mild pain (n=50,60) | 30 | 34
  Day 6; Moderate pain (n=50,60) | 8 | 14
  Day 6; Severe pain (n=50,60) | 2 | 1
  Day 7; No pain (n=50,59) | 8 | 11
  Day 7; Mild pain (n=50,59) | 33 | 34
  Day 7; Moderate pain (n=50,59) | 8 | 12
  Day 7; Severe pain (n=50,59) | 1 | 2
  Day 8; No pain (n=50,59) | 10 | 10
  Day 8; Mild pain (n=50,59) | 29 | 36
  Day 8; Moderate pain (n=50,59) | 11 | 13
  Day 8; Severe pain (n=50,59) | 0 | 0
  Day 9; No pain (n=49,56) | 13 | 10
  Day 9; Mild pain (n=49,56) | 23 | 33
  Day 9; Moderate pain (n=49,56) | 12 | 13
  Day 9; Severe pain (n=49,56) | 1 | 0
  Day 10 or ED; No pain (n=54,60) | 12 | 11
  Day 10 or ED; Mild pain (n=54,60) | 29 | 30
  Day 10 or ED; Moderate pain (n=54,60) | 12 | 18
  Day 10 or ED; Severe pain (n=54,60) | 1 | 1

10. Secondary Outcome: Number of Participants With Total Duration of Pain Per Day in Titration Phase
Description: The participants assessed total painful time in 1 day on a 5-point scale ranging from 0 to 4 where 0 = less than (<) 4 hours, 1 = greater than or equal to (>=) 4 hours to less than 8 hours, 2 = greater than or equal to 8 hours to less than 12 hours, 3 = greater than or equal to 12 hours and 4 = 24 hours (all day).
Time Frame: Day 1 PA, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13 and Day 14 or ED
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Participants
  Day 1 PA; < 4 hours (n=155) | 36
  Day 1 PA; >= 4 to < 8 hours (n=155) | 38
  Day 1 PA; >= 8 to < 12 hours (n=155) | 22
  Day 1 PA; >= 12 hours (n=155) | 24
  Day 1 PA; 24 hours (n=155) | 35
  Day 2; < 4 hours (n=155) | 52
  Day 2; >= 4 to < 8 hours (n=155) | 31
  Day 2; >= 8 to < 12 hours (n=155) | 30
  Day 2; >= 12 hours (n=155) | 17
  Day 2; 24 hours (n=155) | 25
  Day 3; < 4 hours (n=153) | 63
  Day 3; >= 4 to < 8 hours (n=153) | 32
  Day 3; >= 8 to < 12 hours (n=153) | 26
  Day 3; >= 12 hours (n=153) | 12
  Day 3; 24 hours (n=153) | 20
  Day 4; < 4 hours (n=152) | 81
  Day 4; >= 4 to < 8 hours (n=152) | 26
  Day 4; >= 8 to < 12 hours (n=152) | 19
  Day 4; >= 12 hours (n=152) | 13
  Day 4; 24 hours (n=152) | 13
  Day 5; < 4 hours (n=151) | 86
  Day 5; >= 4 to < 8 hours (n=151) | 24
  Day 5; >= 8 to < 12 hours (n=151) | 15
  Day 5; >= 12 hours (n=151) | 14
  Day 5; 24 hours (n=151) | 12
  Day 6; < 4 hours (n=129) | 72
  Day 6; >= 4 to < 8 hours (n=129) | 20
  Day 6; >= 8 to < 12 hours (n=129) | 13
  Day 6; >= 12 hours (n=129) | 12
  Day 6; 24 hours (n=129) | 12
  Day 7; < 4 hours (n=112) | 66
  Day 7; >= 4 to < 8 hours (n=112) | 18
  Day 7; >= 8 to < 12 hours (n=112) | 12
  Day 7; >= 12 hours (n=112) | 7
  Day 7; 24 hours (n=112) | 9
  Day 8; < 4 hours (n=98) | 55
  Day 8; >= 4 to < 8 hours (n=98) | 18
  Day 8; >= 8 to < 12 hours (n=98) | 12
  Day 8; >= 12 hours (n=98) | 6
  Day 8; 24 hours (n=98) | 7
  Day 9; < 4 hours (n=74) | 44
  Day 9; >= 4 to < 8 hours (n=74) | 12
  Day 9; >= 8 to < 12 hours (n=74) | 6
  Day 9; >= 12 hours (n=74) | 4
  Day 9; 24 hours (n=74) | 8
  Day 10; < 4 hours (n=57) | 31
  Day 10; >= 4 to < 8 hours (n=57) | 9
  Day 10; >= 8 to < 12 hours (n=57) | 5
  Day 10; >= 12 hours (n=57) | 4
  Day 10; 24 hours (n=57) | 8
  Day 11; < 4 hours (n=51) | 35
  Day 11; >= 4 to < 8 hours (n=51) | 2
  Day 11; >= 8 to < 12 hours (n=51) | 8
  Day 11; >= 12 hours (n=51) | 1
  Day 11; 24 hours (n=51) | 5
  Day 12; < 4 hours (n=38) | 25
  Day 12; >= 4 to < 8 hours (n=38) | 2
  Day 12; >= 8 to < 12 hours (n=38) | 7
  Day 12; >= 12 hours (n=38) | 2
  Day 12; 24 hours (n=38) | 2
  Day 13; < 4 hours (n=29) | 17
  Day 13; >= 4 to < 8 hours (n=29) | 3
  Day 13; >= 8 to < 12 hours (n=29) | 4
  Day 13; >= 12 hours (n=29) | 3
  Day 13; 24 hours (n=29) | 2
  Day 14 or ED; < 4 hours (n=155) | 107
  Day 14 or ED; >= 4 to < 8 hours (n=155) | 16
  Day 14 or ED; >= 8 to < 12 hours (n=155) | 15
  Day 14 or ED; >= 12 hours (n=155) | 9
  Day 14 or ED; 24 hours (n=155) | 8

11. Secondary Outcome: Number of Participants With Total Duration of Pain Per Day in Double Blind Phase
Description: as for outcome 10
Time Frame: Day 14-End of Titration Phase (ETP), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9 and Day 10 or ED
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
Participants
  ETP; < 4 hours (n=54,60) | 44 | 46
  ETP; >= 4 to < 8 hours (n=54,60) | 5 | 5
  ETP; >= 8 to < 12 hours (n=54,60) | 2 | 7
  ETP; >= 12 hours (n=54,60) | 2 | 1
  ETP; 24 hours (n=54,60) | 1 | 1
  Day 2; < 4 hours (n=54,60) | 40 | 48
  Day 2; >= 4 to < 8 hours (n=54,60) | 6 | 3
  Day 2; >= 8 to < 12 hours (n=54,60) | 4 | 7
  Day 2; >= 12 hours (n=54,60) | 3 | 1
  Day 2; 24 hours (n=54,60) | 1 | 1
  Day 3; < 4 hours (n=54,60) | 42 | 46
  Day 3; >= 4 to < 8 hours (n=54,60) | 5 | 6
  Day 3; >= 8 to < 12 hours (n=54,60) | 4 | 5
  Day 3; >= 12 hours (n=54,60) | 2 | 1
  Day 3; 24 hours (n=54,60) | 1 | 2
  Day 4; < 4 hours (n=54,60) | 39 | 43
  Day 4; >= 4 to < 8 hours (n=54,60) | 7 | 10
  Day 4; >= 8 to < 12 hours (n=54,60) | 4 | 3
  Day 4; >= 12 hours (n=54,60) | 1 | 3
  Day 4; 24 hours (n=54,60) | 3 | 1
  Day 5; < 4 hours (n=51,60) | 37 | 45
  Day 5; >= 4 to < 8 hours (n=51,60) | 7 | 8
  Day 5; >= 8 to < 12 hours (n=51,60) | 3 | 4
  Day 5; >= 12 hours (n=51,60) | 2 | 2
  Day 5; 24 hours (n=51,60) | 2 | 1
  Day 6; < 4 hours (n=50,60) | 35 | 48
  Day 6; >= 4 to < 8 hours (n=50,60) | 8 | 6
  Day 6; >= 8 to < 12 hours (n=50,60) | 2 | 3
  Day 6; >= 12 hours (n=50,60) | 4 | 2
  Day 6; 24 hours (n=50,60) | 1 | 1
  Day 7; < 4 hours (n=50,59) | 36 | 46
  Day 7; >= 4 to < 8 hours (n=50,59) | 9 | 6
  Day 7; >= 8 to < 12 hours (n=50,59) | 2 | 2
  Day 7; >= 12 hours (n=50,59) | 2 | 3
  Day 7; 24 hours (n=50,59) | 1 | 2
  Day 8; < 4 hours (n=50,59) | 38 | 46
  Day 8; >= 4 to < 8 hours (n=50,59) | 7 | 4
  Day 8; >= 8 to < 12 hours (n=50,59) | 4 | 4
  Day 8; >= 12 hours (n=50,59) | 1 | 4
  Day 8; 24 hours (n=50,59) | 0 | 1
  Day 9; < 4 hours (n=49,56) | 37 | 44
  Day 9; >= 4 to < 8 hours (n=49,56) | 7 | 7
  Day 9; >= 8 to < 12 hours (n=49,56) | 4 | 2
  Day 9; >= 12 hours (n=49,56) | 1 | 2
  Day 9; 24 hours (n=49,56) | 0 | 1
  Day 10 or ED; < 4 hours (n=54,60) | 42 | 46
  Day 10 or ED; >= 4 to < 8 hours (n=54,60) | 5 | 6
  Day 10 or ED; >= 8 to < 12 hours (n=54,60) | 6 | 2
  Day 10 or ED; >= 12 hours (n=54,60) | 1 | 5
  Day 10 or ED; 24 hours (n=54,60) | 0 | 1

12. Secondary Outcome: Mean Number of Rescue Doses in Titration Phase
Description: Rescue dose was defined as dose of a fast-acting oral morphine hydrochloride solution or morphine in water solution used in the case of breakthrough pain or lack of analgesic effect.
Time Frame: Day 1 PA, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13 and Day 14 or ED
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Rescue doses
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 155
Rescue doses
  Day 1 PA; (n=155) | 0.3 (0.64)
  Day 2; (n=155) | 0.8 (1.17)
  Day 3; (n=153) | 0.7 (1.03)
  Day 4; (n=152) | 0.6 (1.04)
  Day 5; (n=151) | 0.5 (0.70)
  Day 6; (n=129) | 0.7 (0.93)
  Day 7; (n=112) | 0.5 (0.82)
  Day 8; (n=99) | 0.5 (0.86)
  Day 9; (n=74) | 0.4 (0.66)
  Day 10; (n=57) | 0.4 (0.75)
  Day 11; (n=51) | 0.4 (0.85)
  Day 12; (n=38) | 0.5 (0.83)
  Day 13; (n=29) | 0.3 (0.60)
  Day 14 or ED; (n=155) | 0.2 (0.52)

13. Secondary Outcome: Mean Number of Rescue Doses in Double Blind Phase
Description: as for outcome 12
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9 and Day 10 or ED
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rescue doses
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 60
Rescue doses
  Day 1; (n=54,60) | 0.1 (0.41) | 0.2 (0.44)
  Day 2; (54,60) | 0.3 (0.63) | 0.4 (0.74)
  Day 3; (54,60) | 0.3 (0.70) | 0.4 (0.79)
  Day 4; (54,60) | 0.4 (0.70) | 0.4 (0.79)
  Day 5; (52,60) | 0.3 (0.70) | 0.5 (0.75)
  Day 6; (50,60) | 0.3 (0.71) | 0.6 (0.87)
  Day 7; (50,59) | 0.3 (0.65) | 0.5 (1.04)
  Day 8; (50,59) | 0.5 (0.93) | 0.5 (0.90)
  Day 9; (49,56) | 0.5 (1.10) | 0.5 (0.79)
  Day 10 or ED; (54,60) | 0.2 (0.49) | 0.4 (0.82)

14. Secondary Outcome: Number of Participants With Response Based on Physician's Global Assessment Scale in Titration Phase
Description: The treating physician assessed the therapeutic efficacy of the study drug to control pain on a 2-point scale of effective and ineffective. Number of participants with effective and ineffective therapeutic efficacy with respect to the study drug were reported.
Time Frame: Day 14
Population: The FAS population included all participants who applied at least 1 study drug patch and had 1 VAS assessment performed after application of the study drug. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase)
Number analyzed (Participants) | 154
Participants
  Effective | 145 (0.64)
  Ineffective | 9

15. Secondary Outcome: Number of Participants With Response Based on Physician's Global Assessment Scale in Double Blind Phase
Description: as for outcome 14
Time Frame: Day 10
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Number analyzed (Participants) | 54 | 58
Percentage of participants
  Effective | 53 (0.49) | 58 (0.82)
  Ineffective | 1 | 0

ADVERSE EVENTS:
Time Frame: From signing of the informed consent up to 7 days after the completion or discontinuation of study treatment.
Description: Safety set included 155 participants in Dose Titration Phase, 57 participants in Fentanyl 1-day transdermal patch (Double Blind Phase) and 62 participants in Fentanyl 3-day transdermal patch (Double Blind Phase).
Arm/Group | Fentanyl 1-day Transdermal Patch (Titration Phase) | Fentanyl 1-day Transdermal Patch (Double Blind Phase) | Fentanyl 3-day Transdermal Patch (Double Blind Phase)
Serious Adverse Events (participants affected / at risk) | 14/155 | 9/57 | 11/62
Other Adverse Events (participants affected / at risk) | 128/155 | 47/57 | 48/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl 1-day Transdermal Patch (Titration Phase) (N=155) | Fentanyl 1-day Transdermal Patch (Double Blind Phase) (N=57) | Fentanyl 3-day Transdermal Patch (Double Blind Phase) (N=62)
Sepsis (Infections and infestations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl 1-day Transdermal Patch (Titration Phase) (N=155) | Fentanyl 1-day Transdermal Patch (Double Blind Phase) (N=57) | Fentanyl 3-day Transdermal Patch (Double Blind Phase) (N=62)
Somnolence (Nervous system disorders) | 93 | 34 | 36
Constipation (Gastrointestinal disorders) | 78 | 31 | 36
Diarrhoea (Gastrointestinal disorders) | 11 | 8 | 13
Nausea (Gastrointestinal disorders) | 74 | 32 | 34
Vomiting (Gastrointestinal disorders) | 45 | 17 | 23
Hepatic function abnormal (Hepatobiliary disorders) | 11 | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 6 | 5
Application site erythema (General disorders) | 12 | 7 | 7
Application site pruritus (General disorders) | 10 | 4 | 2
Pyrexia (General disorders) | 12 | 6 | 5
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 5 | 4
Insomnia (Psychiatric disorders) | 0 | 5 | 3
Restlessness (Psychiatric disorders) | 0 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 6
Malaise (General disorders) | 0 | 3 | 2
Blood urea increased (Investigations) | 0 | 3 | 1
Platelet count decreased (Investigations) | 0 | 3 | 1
White blood cell count decreased (Investigations) | 0 | 3 | 4
White blood cell count increased (Investigations) | 0 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the Sponsor requires.